## Bijlage C: toestemmingsformulier deelnemer

## SWITCH - Surgical Ward Innovation: Telemonitored controlled by Healthdot

- Ik heb de informatiebrief gelezen. Ook kon ik vragen stellen. Mijn vragen zijn goed genoeg beantwoord. Ik had genoeg tijd om te beslissen of ik meedoe.
- Ik weet dat meedoen vrijwillig is. Ook weet ik dat ik op ieder moment kan beslissen om toch niet mee te doen met het onderzoek. Of om ermee te stoppen. Ik hoef dan niet te zeggen waarom ik wil stoppen.
- Ik geef de onderzoekers toestemming om mijn aangeleverde gegevens te verzamelen en gebruiken. De onderzoekers doen dit alleen om de onderzoeksvraag van dit onderzoek te beantwoorden en om implementatie te verwezenlijken
- Ik weet dat voor de controle van het onderzoek sommige mensen al mijn gegevens kunnen inzien. Die mensen staan in deze informatiebrief. Ik geef deze mensen toestemming om mijn gegevens in te zien voor deze controle.

Wilt u in de tabel hieronder ja of nee aankruisen?

| Ik geef toestemming om mijn gegevens te bewaren om dit te gebruike ander onderzoek, zoals in de informatiebrief staat. | en voor | Ja □ | Nee□ |
|---|---|---|---|
| Ik geef toestemming om mij eventueel na dit onderzoek te vragen of i meedoen met een vervolgonderzoek. | k wil | Ja □ | Nee□ |
| Contactgegevens | | | |
| Deelnemend arts/onderzoeker: F.M.J.F. Schonck, S.A. Nienhuijs, R.A. | ۹. Bouwma | ın | |
| Vermelding van Bureau Patiëntenbelangen (route 257, bereikbaar via | a telefoonn | ummer | 040 – |
| 239 84 10) voor het melden van klachten | | | |
| Functionaris voor de Gegevensbescherming van de instelling: | | | |
| Naam: Mr. Eline Thijssen-Loeffen E-mailadres: fg@catharinaziekenh | uis.nl. | | |
| Voor meer informatie over uw rechten: | | | |
| F.J.M.F. Schonck, emailadres: <a href="mailto:friso.schonck@catharinaziekenhuis.nl">friso.schonck@catharinaziekenhuis.nl</a> | <u> </u> | | |
| Contactgegevens Catharina ziekenhuis, Michelangelolaan 2, 5623 E. | J Eindhove | n | |
| Telefoonnummer: 040 239 9111, onderzoeksteam chirurgie | | | |
| Ik wil meedoen aan dit onderzoek. | | | |
| Mijn naam is (deelnemer): | | | |
| Handtekening: Datu | m :/_ | _/ | |
| Ik verklaar dat ik deze deelnemer volledig heb geïnformeerd over het | genoemde | onderz | oek. |
| Als er tijdens het onderzoek informatie bekend wordt die de toestemr | ning van de | e deelne | mer |
| zou kunnen beïnvloeden, dan breng ik hem/haar daarvan tijdig op de | hoogte. | | |
| Naam onderzoeker (of diens vertegenwoordiger): | | | |
| Handtekening: Datu | m: / | / | |

De deelnemer krijgt een volledige informatiebrief mee, samen met een versie van het getekende toestemmingsformulier.

nWMO2022.Feb.23 - versie [1.0[23Feb2022]

## DCRF-model proefpersoneninformatie voor nWMO onderzoek- 17-Jan-2021

Deelnemersinformatie